CLINICAL TRIAL: NCT03476252
Title: Diagnostic and Prognostic Utility of Pentraxin 3 in Patients With Acute ST Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Diagnostic and Prognostic Utility of Pentraxin 3 in Patients With Acute STEMI Undergoing Primary PCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina maher hafez, cardiology resident, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PTX3
Record Dates: First submitted 2018-03-12; First posted 2018-03-26 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Stemi group undergoing primary pci
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients (Experimental): ST elevation myocardial infarction
  Interventions: Diagnostic Test: pentraxin 3

INTERVENTIONS:
Diagnostic Test: pentraxin 3 — serum pentraxin 3 level will be assessed using ELISA kits

SUMMARY:
A number of inflammatory markers have been recognized, among which the acute phase reactant C-reactive protein showed a positive correlation with the risk of coronary artery disease in both healthy individuals and those at high risk .

Pentraxin 3 is expressed in atherosclerotic plaques, mainly in macrophages and neutrophils, suggesting that pentraxin 3 may be involved in the progression of atherosclerotic plaque.

* A number of studies demonstrated that increased levels of Pentraxin 3 were associated with the presence and increased severity of coronary artery disease in clinically stable patients undergoing elective coronary angiography .
* Pentraxin 3 levels peak at about 7 h after acute MI, which is substantially earlier than CRP, and thus PTX3 could be a better independent predictor of CHD than CRP .
* Recently, it was shown that the number of the involved vessels, MI type, stent length, culprit lesion, and the need for PCI all had a significant relation with abnormal Pentraxin 3 levels , however, it was not studied with respect of its relation with postprocedural angiographic and clinical outcomes.

We thought to evaluate the role of pentraxin-3 on the preprocedural determinants (Grace score, type of MI, culprit lesion, lesion length, pre-procedural TIMI flow, thrombus burden, severity and complexity of CAD as determined by Syntax score and procedural outcome (post-procedural TIMI flow, no reflow and myocardial perfusion assessed by myocardial blush grade as well as the inhospital clinical outcome of primary Percutaneous coronary intervention in patients with acute ST elevation myocardial infarction.

DETAILED DESCRIPTION:
A number of inflammatory markers have been recognized, among which the acute phase reactant C-reactive protein showed a positive correlation with the risk of coronary artery disease in both healthy individuals and those at high risk .

Pentraxin 3 is expressed in atherosclerotic plaques, mainly in macrophages and neutrophils, suggesting that pentraxin 3 may be involved in the progression of atherosclerotic plaque.

* A number of studies demonstrated that increased levels of Pentraxin 3 were associated with the presence and increased severity of coronary artery disease in clinically stable patients undergoing elective coronary angiography .
* Pentraxin 3 levels peak at about 7 h after acute MI, which is substantially earlier than CRP, and thus PTX3 could be a better independent predictor of CHD than CRP .
* Recently, it was shown that the number of the involved vessels, MI type, stent length, culprit lesion, and the need for PCI all had a significant relation with abnormal Pentraxin 3 levels , however, it was not studied with respect of its relation with postprocedural angiographic and clinical outcomes.

We thought to evaluate the role of pentraxin-3 on the preprocedural determinants (Grace score, type of MI, culprit lesion, lesion length, pre-procedural TIMI flow, thrombus burden, severity and complexity of CAD as determined by Syntax score and procedural outcome (post-procedural TIMI flow, no reflow and myocardial perfusion assessed by myocardial blush grade as well as the inhospital clinical outcome of primary Percutaneous coronary intervention in patients with acute ST elevation myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting to our CCU with acute myocardial infarction (STEMI) undergoing PPCI: chest pain > 30 minutes and ST segment elevation in more than one lead, include the definition of MI with a reference: Third universal definition of MI.

Exclusion Criteria:

1. Patients complicated with an infectious disease on admission, active systemic inflammatory disease or chronic inflammatory disease(systemic lupus ,rheumatoid arthritis ,etc).
2. Immune system disease or glucocorticoid therapy.
3. Patients with history of cancer
4. Patients of chronic kidney disease
5. Patients on regular treatments with statins
6. Patients of valvular heart disease, atrial fibrillation (positive relation was proved by previous studies), heart failure and/or cardiogenic shock.
7. Patients underwent previous elective pci or previous CABG.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Measuring relation between pentraxin 3 level and severity of coronary artery disease | two years
  Number of st elevation patients will be investigated before primary percutaneous coronary intervention by measuring serum pentraxin 3 level aiming for good clinical short term outcomes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Knoflach M, Kiechl S, Mantovani A, Cuccovillo I, Bottazzi B, Xu Q, Xiao Q, Gasperi A, Mayr A, Kehrer M, Willeit J, Wick G. Pentraxin-3 as a marker of advanced atherosclerosis results from the Bruneck, ARMY and ARFY Studies. PLoS One. 2012;7(2):e31474. doi: 10.1371/journal.pone.0031474. Epub 2012 Feb 3. PMID 22319633